Title: Adherence to Guidelines VAccination in Type 1 Dlabetes Mellitus Patients (AVADI-1).

NCT03478254 Unique Protocol ID: C-127.

Date: July 15th 2017

## Statistical analysis:

All adult patients suffering T1DM from our electronic database were contacted. We assumed a 15% dropout rate.

Estimated prevalence of T1DM in our area is 0.3%.

Quantitative variables are expressed as means and standard deviation (SD); qualitative variables are presented as total numbers and per-centages.

A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test.

The influence of age, diabetes duration, diabetes complications, glycemic control, type of insulin treatment and health professional job dedication were determined by calculating odds ratios (OR) with a 95% confidence interval (CI).

Multiple regression was used to search for significant predictors elements of studied vaccinations. Significance was taken at P < 0.05.

Analyses were performed with IBM SPSS software version 21.0 for Windows (SPSS Inc., Chicago, IL).